CLINICAL TRIAL: NCT02078453
Title: CARies DEtection in Children - Impact of the Radiographic Examination on Diagnosis and Treatment Decision of Caries Lesions in Primary Teeth
Brief Title: Impact of the Radiographic Examination on Diagnosis and Treatment Decision of Caries Lesions in Primary Teeth
Acronym: CARDEC-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Fausto Medeiros Mendes, Associate professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: CARDEC-01
Record Dates: First submitted 2014-02-25; First posted 2014-03-05 (Estimated); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Dental Caries; Teeth Loss; Quality of Life
Keywords: Dental caries; Diagnosis; Visual inspection; Radiographic examination
MeSH Terms: conditions — Dental Caries; Anodontia; Disease | interventions — Dental Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visual inspection (Active Comparator): Dental treatment performed according to the caries diagnosis obtained with visual inspection performed alone
  Interventions: Procedure: Dental treatment
- Radiographic examination (Experimental): Dental treatment performed according to the caries diagnosis obtained with visual inspection and additional radiographic method.
  Interventions: Procedure: Dental treatment

INTERVENTIONS:
Procedure: Dental treatment — Dental treatment of all dental needs present in the children related or not to the dental caries.

SUMMARY:
Radiographs have been used to aid dentists in detecting the presence of cavities in the deciduous teeth of children. This procedure is globally recommended because the conventional clinical examination usually overlooks some cavities. However, the real benefit of performing dental radiographs for this purpose is still unclear. Besides the hazards of ionizing radiation, the radiographs could provoke overtreatment of the children; hence, dentists would tend to restore more teeth than would be really necessary. Nowadays, it is preferable to overlook some cavities than treat the teeth unnecessarily. Therefore, the investigators aimed to perform this study to compare two different strategies for detecting cavities in deciduous teeth of children: one based on clinical examination performed alone and other using radiographs adjunct to the clinical examination. To compare these strategies, the investigators will consider outcomes related to children's health and welfare.

DETAILED DESCRIPTION:
Despite most clinical guidelines throughout the world indicate that the clinicians take two bitewings for detecting caries lesions in primary molars of asymptomatic children, the evidence for this recommendation is based in cross-sectional studies performed in laboratorial setting or using convenience samples. The benefits and impact of performing radiographs on diagnosis and treatment decision of caries lesions in primary teeth, considering relevant outcomes for the patients, have not been evaluated yet. Thus, the aim of this study will be to evaluate the impact of performing radiographic examination for detecting caries lesions in primary teeth compared with the visual inspection performed alone, considering different outcomes related to the validity and children's health and welfare. For this, three different studies will be carried out according the following specific aims: (1) to evaluate the validity of radiographic examination adjunct to the visual inspection in detecting proximal caries lesions in primary molars in children with low and high caries experience through a cross-sectional design; (2) to evaluate the impact of radiographic examination adjunct to the visual inspection on the diagnostic and treatment decision of caries lesions in primary teeth in a before and after study; and (3) to evaluate the impact of radiographic examination adjunct to the visual inspection for detecting caries lesions in primary teeth on operative needs in the follow-ups and impact of oral health on the quality of life through a randomized clinical trial. To reach these objectives, 250 children aged 3 to 6 years who looked for dental treatment in our dental school will be randomly allocated in two groups according to the diagnostic strategy used for caries detection: visual inspection performed alone (control group) or visual inspection associated to radiographic examination (experimental group). After elaboration of treatment decision plan for two examiners, the children will be treated and followed-up for 2 years, with evaluations after 12 and 24 months after the ingress of the children in the study. The primary outcome will be the number of dental surfaces with dental treatment need in the follow-up, considering the aim (3). Then, children allocated in the control group will be reevaluated using radiographic examination, and the performance of two strategies for detecting proximal caries lesions will be evaluated, using temporary separation with orthodontic rubbers for one week as reference standard method. Moreover, a new treatment plan will be performed and compared with the treatment plan based on visual inspection alone. These two parts of the research will be carried out to reach the aims (1) and (2), respectively. Our working hypothesis is that the radiographic examination would actually exert little influence on outcomes related to the validity and children's health and welfare, and that visual inspection would be enough as diagnostic strategy for caries detection in primary teeth.

ELIGIBILITY:
Inclusion Criteria:

* Children who sought dental treatment in our dental school (School of Dentistry, University of Sao Paulo, Sao Paulo, Brazil)
* Children aged 3 to 6 years
* Children with al least one primary molar in the mouth.

Exclusion Criteria:

* Children whose parents refuse to participate of the research
* Children presenting behavior problems during the treatment.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 252 (Actual)
Dates: Start 2014-03; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Number of dental surfaces with operative treatment needs | 24 months
  The number of dental surfaces with operative treatment needs after the follow-ups will be composed by number of surfaces with new caries lesions; number of restored surfaces with necessity of replacement; tooth with pain episode and/or necessity of endodontic treatment and tooth indicated for extraction.

SECONDARY OUTCOMES:
Number of surfaces with new caries lesions | 24 months
  Dental surfaces presenting caries lesions in the foloow-up examinations that require operative treatment.
Number of restored surfaces with necessity of replacement | 24 months
  Number of restored dental surfaces that requires repair or replacement.
Episodes of dental pain and/or primary teeth with pulpal involvement | 24 months
  Number of primary teeth that presented pain episodes or that require endodontic treatment in the follow-up examinations
Primary teeth indicated for extraction due to caries | 24 months
  Number of primary teeth indicated for extraction due caries involvment.

OTHER OUTCOMES:
Impact of Oral Health on quality of life | 24 months
  Impact of Oral Health on quality of life of the children participants in the study, measured by a validated questionnaire (ECOHIS)

CONTACTS AND LOCATIONS:
Overall Officials: Fausto M Mendes, PhD, Principal Investigator — School of Dentistry, University of Sao Paulo
Locations (1):
- School of Dentistry, University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Novaes TF, Pontes LRA, Freitas JG, Acosta CP, Andrade KCE, Guedes RS, Ardenghi TM, Imparato JCP, Braga MM, Raggio DP, Mendes FM; CARDEC collaborative group. Responsiveness of the Early Childhood Oral Health Impact Scale (ECOHIS) is related to dental treatment complexity. Health Qual Life Outcomes. 2017 Sep 20;15(1):182. doi: 10.1186/s12955-017-0756-z. PMID 28931398
- [Result] Pontes LRA, Novaes TF, Lara JS, Moro BLP, Gimenez T, Raggio DP, Braga MM, Mendes FM. Impact of the radiographic method on treatment decisions related to dental caries in primary molars: a before-after study. Clin Oral Investig. 2019 Nov;23(11):4075-4081. doi: 10.1007/s00784-019-02844-w. Epub 2019 Feb 18. PMID 30778687
- [Derived] Freitas JG, Pontes LRA, Acosta CP, Novaes TF, Lara JS, Gimenez T, Ardenghi TM, Braga MM, Raggio DP, Mendes FM; CARDEC collaborative group. Influence of two caries detection strategies on the quality of life of preschool children: An analysis of secondary outcomes of a 2-Year randomized clinical trial. Community Dent Oral Epidemiol. 2023 Oct;51(5):804-812. doi: 10.1111/cdoe.12765. Epub 2022 Jun 7. PMID 35670271
- [Derived] Pontes LRA, Lara JS, Novaes TF, Freitas JG, Gimenez T, Moro BLP, Maia HCM, Imparato JCP, Braga MM, Raggio DP, Mendes FM; CARDEC collaborative group. Negligible therapeutic impact, false-positives, overdiagnosis and lead-time are the reasons why radiographs bring more harm than benefits in the caries diagnosis of preschool children. BMC Oral Health. 2021 Mar 31;21(1):168. doi: 10.1186/s12903-021-01528-w. PMID 33789655
- [Derived] Pontes LRA, Novaes TF, Lara JS, Gimenez T, Moro BLP, Camargo LB, Michel-Crosato E, Pannuti CM, Raggio DP, Braga MM, Mendes FM. Impact of visual inspection and radiographs for caries detection in children through a 2-year randomized clinical trial: The Caries Detection in Children-1 study. J Am Dent Assoc. 2020 Jun;151(6):407-415.e1. doi: 10.1016/j.adaj.2020.02.008. PMID 32450979
- [Derived] Mendes FM, Pontes LR, Gimenez T, Lara JS, de Camargo LB, Michel-Crosato E, Pannuti CM, Raggio DP, Braga MM, Novaes TF; CARDEC Collaborative Group. Impact of the radiographic examination on diagnosis and treatment decision of caries lesions in primary teeth--the Caries Detection in Children (CARDEC-01) trial: study protocol for a randomized controlled trial. Trials. 2016 Feb 9;17:69. doi: 10.1186/s13063-016-1196-5. PMID 26857821